CLINICAL TRIAL: NCT06994676
Title: CROSSCHECK-001: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate Safety, Tolerability, and Clinical Activity of CBX-250 in Participants With Relapsed or Refractory Acute Myeloid Leukemia, High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: A Study of CBX-250 in Participants With Acute Myeloid Leukemia, High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Acronym: CROSSCHECK-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Crossbow Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBX-250-001
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: High-risk Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia (CMML); AML - Acute Myeloid Leukemia
Keywords: AML; HR-MDS; CMML; acute leukemia; CBX-250; CBX-250-001; CROSSCHECK; CROSSCHECK-001; Crossbow
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBX-250 (Experimental): subcutaneous CBX-250
  Interventions: Drug: CBX-250

INTERVENTIONS:
Drug: CBX-250 — subcutaneous CBX-250

SUMMARY:
Study CBX-250-001 is a Phase 1, open-label, dose-escalation study of CBX-250 in participants with relapsed/refractory AML, HR-MDS and CMML. Participants aged ≥ 12 years are planned to be enrolled. CBX-250 will initially be investigated on a fixed step-up dosing schedule. CBX-250 will be administered subcutaneously in 28-day cycles, with the first study drug dose administered on Cycle 1, Day 1. Cycle 1 will consist of a priming phase over 7 days, and a target phase over 28 days. Participants will continue CBX-250 until progressive disease (PD) or unacceptable toxicity. All subsequent treatment cycles will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Dose Escalation: Male or female participants aged ≥18 years.
2. Backfill Cohorts: Male or female participants aged ≥12 years for whom no curative treatment options, including transplantation, are available.

   Diagnosis & Disease Characteristics
3. Participants with histological confirmation of advanced hematologic malignancy including:

   1. R/R AML, as defined by standardized criteria (e.g., European LeukemiaNet criteria [Dohner 2022]; after standard of care therapy. Participants with persistent leukemia after initial therapy or with recurrence of leukemia at any time after achieving a response during or after the course of treatment (including HSCT) are eligible.
   2. R/R HR-MDS or very high risk MDS as per the Revised International Prognostic Scoring System (IPSS-R; Greenberg 2012) or Molecular International Prognostic Scoring System (IPPS-M, Bernard 2022) who are resistant or refractory to 4-6 cycles of hypomethylating agents (HMA; decitabine or azacitidine).
   3. R/R CMML who are resistant or refractory to 4-6 cycles of hypomethylating agents (HMA; decitabine or azacitidine).
4. White blood cells must be below 25,000/µL at time of enrollment. Participants may receive cytoreduction prior to enrollment.
5. Historical documented evidence of HLA-A*02:01 allele positivity.

   Performance Level
6. ECOG PS score 0-1 (if aged ≥18 years); Karnofsky Performance Scale of ≥70 (if aged ≥16 years and <18 years); Lansky PS of ≥70 (if aged <16 years).

   Prior Therapy
7. Any prior treatment-related toxicities resolved to ≤Grade 1 prior to enrollment, with the exception of ≤Grade 2 alopecia.
8. Radiation Therapy: At least 60 days from prior total body irradiation, craniospinal radiation and/or ≥50% radiation of the pelvis, or at least 14 days from local palliative radiation therapy (small port).
9. Stem Cell Infusion: At least 60 days must have elapsed from HSCT and at least 4 weeks (from first dose) must have elapsed from donor lymphocyte infusion without conditioning.
10. Immunotherapy: At least 42 days since prior immunotherapy, including tumor vaccines and checkpoint inhibitors, and at least 21 days since receipt of chimeric antigen receptor therapy.
11. Anti-Leukemia Therapy: At least 14 days since the completion of anti-leukemic therapy (for example, but not limited to, small molecule or cytotoxic/myelosuppressive therapy), with the following exceptions:

    * Hydroxyurea for cytoreduction can be initiated without restriction related to timing of study entry. Hydroxyurea for cytoreduction can be continued concomitantly with CBX-250, with Study Responsible Physician approval.
    * Intrathecal chemotherapy at the time of diagnostic lumbar puncture at least 24 hours prior to the start of CBX-250 and may continue prophylactic intrathecal chemotherapy beginning in Cycle 2, at the treating physician's discretion.
12. Hematopoietic Growth Factors: At least 7 days since the completion of therapy with short-acting hematopoietic growth factors and 14 days with long-acting growth factors.
13. Biologics (e.g. monoclonal antibody therapy): At least 28 days or 5 half-lives, whichever is shorter, have elapsed since the completion of therapy with a biologic agent. Any AE related to prior biologic treatment must be resolved to baseline severity or ≤Grade 1.
14. Steroids: At least 7 days since systemic glucocorticoid therapy, unless receiving physiologic dosing (equivalent to ≤10 mg prednisone daily) or cytoreductive therapy. Cytoreductive therapy must have approval of the Study Responsible Physician.

    Adequate Organ Function Requirements within 10 Days of Treatment Initiation
15. Estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2 based on local institutional practice for age-appropriate determination (eg, Schwartz formula for pediatric participants or Cockcroft-Gault formula for adults).

    1. Participants ≥18 years: glomerular filtration rate ≥45 mL/min
    2. Participants <18 years: ≥45 mL/min x (participant's body surface area m2/1.73) • Adequate liver function defined as:

       * Total bilirubin <1.5 × the upper limit of normal (ULN) for age or normal conjugated bilirubin, or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in participants with well documented Gilbert's syndrome or hemolysis or who require regular blood transfusions.
       * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 × ULN (unless attributed to leukemic involvement with discussion with the Study Responsible Physician).

    Sex and Contraceptive/Barrier Requirements
16. If a female of childbearing potential, willing to use a highly effective method of contraception or double barrier method from the time of enrollment through 120 days following the last study drug dose.
17. If male of childbearing potential, agrees to use barrier contraception from the time of enrollment through 120 days following the last study drug dose.

    Informed Consent
18. Participant or participant's health care proxy is able and willing to provide written informed consent and able to follow study instructions.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Diagnosis

1. Previous CTSG targeted therapy or treatment with any pMHC T-cell engager.
2. Isolated extramedullary relapse.
3. Active central nervous system (CNS) disease. Participants with prior CNS history can be enrolled if the participant has a negative lumbar puncture following completion of intrathecal chemotherapy).

   Infection
4. Known HIV infection.
5. Active hepatitis B infection (participants with documented clearance following treatment are allowed).
6. Active hepatitis C infection (participants with documented clearance following treatment are allowed).

   Pregnancy and Breastfeeding
7. Pregnant or nursing women: Negative serum pregnancy tests are required during Screening and a negative serum or urine pregnancy test is required within 72 hours prior to receiving the first study drug administration, in females of childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Concurrent Conditions
8. Cardiac Disease:

   * Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class >II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
   * QTc using Fridericia's correction (QTcF) >480 msec
9. Graft-Versus-Host Disease (GVHD): Active acute or chronic GVHD requiring systemic treatment with immunosuppressive medication. Participants may be on physiological doses of steroids.
10. Concurrent malignancy in the previous 2 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ, melanoma in situ) treated with potentially curative therapy. Concurrent malignancy must be in CR or no evidence of disease (NED) during this timeframe.
11. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate.

    Concomitant Medications and Interventions
12. Any commercially available or investigational anti-leukemic therapy other than CBX-250, with the following exceptions:

    • Intrathecal chemotherapy for CNS prophylaxis is permitted after C1 is complete, at the treating physician's discretion.
13. Participation in another therapeutic interventional clinical study in which an investigational agent was administered within 14 days or 5-halflives, whichever is shorter, of starting CBX-250. Participants may continue with non-interventional follow-up from previous clinical studies.
14. Any concurrent systemic treatment to prevent GVHD. Topical treatments for GVHD are permitted.
15. Known allergy or sensitivity to study drug, including excipients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To determine the safety, tolerability, RP2D, or MTD if different, and dosing regimen of CBX-250. | Until the end of study (approximately 24 months)
  Frequency and type of DLT
To determine the safety, tolerability, RP2D, or MTD if different, and dosing regimen of CBX-250. | Until the end of study (approximately 24 months)
  Frequency, duration, and severity of TEAEs, TRAEs, AESIs, and SAEs
To determine the safety, tolerability, RP2D, or MTD if different, and dosing regimen of CBX-250. | Until the end of study (approximately 24 months)
  Frequency and severity of CRS AEs
To determine the safety, tolerability, RP2D, or MTD if different, and dosing regimen of CBX-250. | Until the end of study (approximately 24 months)
  Drug withdrawals, drug interruptions, or dose reductions due to adverse events
To determine the safety, tolerability, RP2D, or MTD if different, and dosing regimen of CBX-250. | Until the end of study (approximately 24 months)
  Incidence/shifts of clinical laboratory abnormalities

SECONDARY OUTCOMES:
AUC0-t (first dose and at steady state) | Approximately 1 year
  Area under the plasma concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of CBX-250 and relevant metabolites
Cmax | Approximately 1 year
  Maximum plasma concentration (Cmax) of CBX-250 and relevant metabolites
Tmax | Approximately 1 year
  Time to observed maximum plasma concentration of CBX-250 and relevant metabolites
ADAs | Approximately 1 year
  Incidence and severity of anti-drug antibodies
ORR | Approximately 1 year
  To assess the overall response rate (ORR) of CBX-250
CR+CRh rate in AML | Approximately 1 year
  To assess the complete remission (CR) and complete remission with partial hematologic recovery (CRh) rate
EFS | Approximately 3 years
  To assess the event free survival (EFS) of CBX-250
OS | Approximately 3 years
  To assess overall survival (OS) of CBX-250
DOR | Approximately 3 years
  To assess the duration of response (DOR) of CBX-250
CRc rate in AML | Approximately 3 years
  To assess the composite definition of complete remission (CRc) rate
Remission rate in HR-MDS | Approximately 1 year
  Remission rate as defined by Zeidan 2023: CR, CR equivalent, partial remission (PR), CRL (CRuni and CRbi), CRh, Hematologic improvement (HI)
PFS | Approximately 3 years
  To assess the progression free survival (PFS) of CBX-250
CR+CRh rate in HR-MDS | Approximately 1 year
  CR+ CR equivalent+ CRL + CRh
Transfusion independence | Approximately 3 years
  Any transfusion-free period lasting for at least 56 consecutive days, during which the participant is either on CBX-250 therapy or after cessation of CBX-250 therapy but prior to the start of new therapy
To assess the preliminary anti-leukemic activity of CBX-250 in participants with CMML | Approximately 1 year.
  Proportion of participants achieving complete response (CR), complete cytogenetic remission, partial response (PR), marrow response, and clinical benefit according to the 2015 International Consortium Proposal of Uniform Response Criteria for Myelodysplastic Syndromes (MDS)/Myeloproliferative Neoplasms (MPN).

CONTACTS AND LOCATIONS:
Overall Officials: Briggs Morrison, MD, Study Chair — Crossbow Therapeutics, Inc.
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Cancer Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the results of this study may be presented at scientific meetings and/or published in a peer reviewed scientific or medical journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after publication
Access Criteria: Requests to be reviewed on an individual basis by Crossbow Therapeutics, Inc.